CLINICAL TRIAL: NCT02192619
Title: National Acute Promyelocytic Leukemia (APL) Observational Study NAPOLEON-Registry of the German AML Intergroup
Status: Recruiting | Type: Observational
Sponsor: Gesellschaft fur Medizinische Innovation - Hamatologie und Onkologie mbH (Other)
Responsible Party: Sponsor
Other Study IDs: NAPOLEON-Registry
Record Dates: First submitted 2014-07-11; First posted 2014-07-17 (Estimated); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Newly-diagnosed APL (de Novo or Therapy-related); Relapsed APL
Keywords: APL; acute promyelocytic leukemia; AML M3
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- observational
  Interventions: Other: observational

INTERVENTIONS:
Other: observational

SUMMARY:
The registry aims to document epidemiologic data, treatment and long-term outcome as well as quality of life of patients with APL. Additionally, a biobanking project for further translational studies is integrated.

Prospective population-based non-interventional and non-randomized multicenter registry.

DETAILED DESCRIPTION:
* collection of epidemiological data for APL: age distribution, prognostic factors, distribution of subgroups, incidence
* documentation of efficacy and safety of the first line and salvage therapy in APL including
* documentation of minimal residual disease (MRD)
* correlation of clinical outcomes with chosen therapy
* collection and evaluation of quality of life
* validation of published prognostic factors / new potential prognostic factors
* acquisition of bone marrow, peripheral blood and buccal swab samples for biobanking and translational studies under the umbrella of the specific study-group biobanking concepts

ELIGIBILITY:
Inclusion Criteria:

* newly-diagnosed APL (either de novo or therapy-related), within 12 months of diagnosis
* or relapsed APL, within 12 months of diagnosis of relapse

  1. confirmed by the presence of the translocation t(15; 17)
  2. and / or confirmed by the detection of the fusion transcript of PML/RARa

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly-diagnosed or relapsed APL (de novo or therapy-related) who require a therapeutic intervention according to their disease state are the study population within this registry.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
epidemiological parameters | yearly follow up for 5 years
diagnostic quality indicators | yearly follow up for 5 years
type of therapy | yearly follow up for 5 years
response, recurrence and time of death and resulting outcomes RFS and OS | yearly follow up for 5 years

SECONDARY OUTCOMES:
complete remission (CR) and CRm | yearly follow up for 5 years
treatment related mortality (TRM) | yearly follow up for 5 years
cumulative incidence of relapse (CIR) | yearly follow up for 5 years
grade IV toxicities | yearly follow up for 5 years
quality of life (QoL): EORTC QLQ-C30 | yearly follow up for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard F. Schlenk, Prof. Dr., Principal Investigator — Universitätsklinikum Ulm, for the AML-SG group; Eva Lengfelder, PD Dr., Principal Investigator — Universitätsklinikum Mannheim; Dietger Niederwieser, Prof. Dr., Principal Investigator — Universitätsklinikum Leipzig
Locations (1):
- Prof. Dr. U. Platzbecker, Dresden, Germany

REFERENCES:
- [Derived] Kayser S, Schlenk RF, Lebon D, Carre M, Gotze KS, Stolzel F, Berceanu A, Schafer-Eckart K, Peterlin P, Hicheri Y, Rahme R, Raffoux E, Chermat F, Krause SW, Aulitzky WE, Rigaudeau S, Noppeney R, Berthon C, Gorner M, Jost E, Carassou P, Keller U, Orvain C, Braun T, Saillard C, Arar A, Kunzmann V, Wemeau M, De Wit M, Niemann D, Bonmati C, Schwanen C, Abraham J, Aljijakli A, Haiat S, Kramer A, Reichle A, Gnadler M, Willekens C, Spiekermann K, Hiddemann W, Muller-Tidow C, Thiede C, Rollig C, Serve H, Bornhauser M, Baldus CD, Lengfelder E, Fenaux P, Platzbecker U, Ades L. Characteristics and outcome of patients with low-/intermediate-risk acute promyelocytic leukemia treated with arsenic trioxide: an international collaborative study. Haematologica. 2021 Dec 1;106(12):3100-3106. doi: 10.3324/haematol.2021.278722. PMID 34047178
- See also: Related Info — http://www.gmiho.de/
- See also: Related Info — http://www.aml-germany.com/